CLINICAL TRIAL: NCT01037478
Title: A Phase 2 Proof of Concept Study to Evaluate the Efficacy, Safety and Pharmacokinetics of the HDAC Inhibitor 4SC-201 in Patients With Relapsed or Refractory Hodgkin's Lymphoma
Brief Title: Resminostat (4SC-201) in Relapsed or Refractory Hodgkin's Lymphoma
Acronym: SAPHIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 4SC AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4SC-201-2-2009
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; HDAC; 4SC-201; Resminostat; Phase II
MeSH Terms: conditions — Hodgkin Disease | interventions — resminostat

ARMS (1):
- Resminostat (4SC-201) (Experimental): oral administration
  Interventions: Drug: Resminostat (4SC-201)

INTERVENTIONS:
Drug: Resminostat (4SC-201) — oral administration

SUMMARY:
The purpose of this study is to determine whether Resminostat (4SC-201) is effective and safe in the treatment of relapsed or refractory Hodgkin's Lymphoma.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients must have histological or cytological evidence of Hodgkin's Lymphoma (all subtypes are acceptable)
* Patients must have relapsed or refractory Hodgkin's Lymphoma (HL) defined as relapse following initial therapy or lack of response to first line therapy and treatment with second-line (salvage therapy). Patients may have also undergone high-dose chemotherapy with autologous stem cell transplantation at least 12 weeks prior to study entry
* Patients must have measurable anatomical disease present on CT scan
* Patients must have an ECOG Performance Score of 0, 1 or 2

Main Exclusion Criteria:

* Patients who have received previous treatment with an HDAC inhibitor
* Patients who have undergone allogeneic hematopoietic stem cell transplantation
* Patients with known or suspected involvement of the CNS by HL
* Patients treated with agents known to prolong the QT interval or with a confirmed QTcF > 450 msec
* Patients with a history of other malignancies unless having undergone definitive treatment more than 5 years prior to entry into the study and without evidence of recurrent malignant disease, excluding patients with basal cell carcinoma of the skin; superficial carcinoma of the bladder; carcinoma of the prostate with a current PSA < 0.1 ng/ml; or cervical intraepithelial neoplasia
* Patients with a history of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory or inflammatory illness that could preclude their participation in the trial, pose an undue medical hazard or interfere with the interpretation of the trial results, including, but not limited to, patients with congestive heart failure (NYHA Class 3 or 4); unstable angina; cardiac arrhythmia; recent (within the preceding 6 months) myocardial infarction or stroke; hypertension requiring > 2 medications for adequate control; diabetes mellitus with > 2 episodes of ketoacidosis in the preceding 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determination of the best overall objective response rate (ORR) based on IWG criteria of Resminostat (4SC-201) in patients with refractory or relapsed Hodgkin's Lymphoma. | 12 weeks

SECONDARY OUTCOMES:
Investigation of the safety and tolerability of repeated oral doses of Resminostat (4SC-201) | 12 weeks
Assessment of the overall survival (OS) | 12 weeks
Determination of progression free survival (PFS), including radiological and symptomatic progression | 12 weeks
Determination of time to progression (TTP), including objective and symptomatic progression | 12 weeks
Determination of duration of response (DOR) | 12 weeks
Assessment of the pharmacokinetics of Resminostat (4SC-201) after oral dosing | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan Walewski, Prof., Principal Investigator — Instytut im. Marii Skłodowskiej-Curie, Centrum Onkologii, Warsaw, Poland
Locations (10):
- Czechia (3):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice Hradec Kralové, Hradec Kralové
  - Fakultní nemocnice Kralovske Vinohrady, Prague
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Nr.1 w Poznaniu, Poznan
  - Instytut im. Marii Sklodowskiej-Curie, Centrum Onkologii, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr.1 we Wroclawiu, Wroclaw
- Romania (2):
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Coltea, Bucharest